CLINICAL TRIAL: NCT04553588
Title: Implementation of a Program for Safe Medication Disposal in a Perioperative Unit: A Response to the Opioid Crisis
Brief Title: Effect of an Opioid Disposal Pouch Versus Usual Care on Post Discharge Disposal of Unused Medication
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Antoinette Zito, Perioperative Educator, Office of Nursing Education and Professional Development, Principal Investigator, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 17-801
Record Dates: First submitted 2020-09-07; First posted 2020-09-17 (Actual); Last update posted 2020-09-17 (Actual); Status verified 2020-09

CONDITIONS: Drug Prescriptions
Keywords: opioid misuse; disposal; disposal pouch; postoperative surgery
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: Two group design; patients randomized to receive usual postoperative care after discharge or usual postoperative care plus a disposal pouch to safely eliminate opioid medication no longer needed
Who Masked: Care Provider
Masking Description: Care provider did not receive communication regarding group assignment; patients allocated to the intervention group received a disposal pouch prior to discharge and after physician discharge orders were finalized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Opioid Disposal Pouch (Active Comparator): an opioid disposal pouch to inactivate and dispose of unused opioid medication within the first 30 days after surgery
  Interventions: Other: Disposal pouch
- Usual Care (No Intervention): usual medication disposal includes multiple options as desired by patient; for example, flushing down toilet, giving to local pharmacist, giving to police department etc.

INTERVENTIONS:
Other: Disposal pouch — Medication Disposal Pouch
  Other Names: Medsaway Pouch
  Arms: Opioid Disposal Pouch

SUMMARY:
The purpose of the study is to determine if opioid disposal bags/pouches are an effective method for disposing of unused opioid medications postoperatively

DETAILED DESCRIPTION:
Opioids are dispensed regularly to manage postoperative pain in patients undergoing surgery in hospitals and same day surgery centers. There has been a rise in the number of opioid misuse and overdoses nationally, with Ohio ranked first in the nation for drug overdose deaths in 2014 and Cuyahoga County leading the state with 666 overdose deaths in 2016(ref) As health care providers, it is our responsibility to respond to this epidemic. One measure to address this is to reduce the number of unused prescription opioids that remain in patients' possession when they no longer need them. (ref) Doing so will maximize safety by decreasing the availability of unused opioids. The purpose of this study is to determine if a product that deactivates opioids will be used as designed after oral opioid medication is no longer needed. The design of this study is a quality initiative project using a randomized control design. The setting is a surgery center in a suburban hospital in Cuyahoga County. The population is all adult surgery center patients that are prescribed opioids postoperatively who are discharged the same day. In addition to usual care, a medication disposal bag with instructions on how to use will be given to the patient prior to discharge. The patient will be called 30-45 days post discharge. The data will be collected on a case report form that will include information about disposal and information obtained from the patients medical record.

ELIGIBILITY:
Inclusion Criteria

* Adults (>18 years)
* Scheduled to go home on the day of surgery
* Received a prescription for opioids
* Willing to provide a telephone number and receive a phone call 30 days after surgery

Exclusion Criteria

* Moderate to severe cognitive decline requiring caregiver support
* Not able to speak or understand English (instructions only available in English)
* Behavioral health diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 313 (Actual)
Dates: Start 2017-07-15 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2020-02-27 (Actual)

PRIMARY OUTCOMES:
Rate of Disposal of Unused Opioid Medication | 30 days postoperatively
  rate of patient reported unused oral opioid medication disposal between groups

SECONDARY OUTCOMES:
Odds of disposal pouch use after adjusting for group assignment | 30 days postoperatively
  Odds of disposal pouch use after adjusting for group assignment (usual care versus disposal pouch group)
Odds of disposal pouch use after adjusting for pain level on the worst day of postoperative pain | 30 days postoperatively
  Odds of disposal pouch use after adjusting for pain level on the worst day of postoperative pain
Odds of disposal pouch use after adjusting for preoperative opioid use | 30 days postoperatively
  Odds of disposal pouch use after adjusting for preoperative opioid use
Odds of disposal pouch use after adjusting for race | 30 days postoperatively
  Odds of disposal pouch use after adjusting for race
Odds of disposal pouch use after adjusting for gender | 30 days postoperatively
  Odds of disposal pouch use after adjusting for gender
Odds of disposal pouch use after adjusting for surgical procedure type | 30 days postoperatively
  Odds of disposal pouch use after adjusting for surgical procedure type
Odds of disposal pouch use after adjusting for insurance type | 30 days
  Odds of disposal pouch use after adjusting for insurance type

CONTACTS AND LOCATIONS:
Overall Officials: Zito Antoinette, MSN, Principal Investigator — Cleveland Clinic Health System
Locations (1):
- Cleveland Clinic Health System, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No